CLINICAL TRIAL: NCT01187849
Title: Metformin to Prevent Metabolic Complications in Glucocorticoid Excess
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: EKBB 245/09
Record Dates: First submitted 2010-08-23; First posted 2010-08-24 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Patients With Glucocorticoid Treatment
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin (Active Comparator)
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — Volunteers will be given Metformin or placebo for 1 month, once daily.
  Arms: Metformin
Drug: Placebo — Volunteers will be given Metformin or placebo for 1 month, once daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate if a treatment with metformin compared to placebo reduces metabolic side-effects in patients with glucocorticoid treatment over three months time.

ELIGIBILITY:
Inclusion Criteria:

* Glucocorticoid treatment for ≥ 3 months with a prednisone dose of ≥ 7.5mg/d or equivalent glucocorticoid

Exclusion Criteria:

* Refusal of informed consent
* Prior therapy with metformin during the last 6 month
* Preexisting diabetes
* Pregnancy or current malignancy
* Renal insufficiency with a creatinine clearance lower than 30ml/min

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2010-08; Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
2 hours glucose level after a standardized 75g oral glucose tolerance test (OGTT) | 0 months, 3 months

SECONDARY OUTCOMES:
homeostasis model assessment (HOMA)-index | 0 months, 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Mirjam Christ-Crain, MD, Prof., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No